CLINICAL TRIAL: NCT00077662
Title: A Prospective, Observational Study in Patients With Late-Onset Pompe Disease
Status: Completed | Type: Observational
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Other Study IDs: AGLU02303; "LOPOS"
Record Dates: First submitted 2004-02-10; First posted 2004-02-12 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Glycogen Storage Disease Type II
Keywords: Pompe Disease; Glycogen Storage Disease Type II; GSD-II; Acid Maltase Deficiency Disease; Glycogenosis 2
MeSH Terms: conditions — Glycogen Storage Disease Type II

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Pompe disease (also known as glycogen storage disease type II, "GSD-II") is caused by a deficiency of a critical enzyme in the body called acid alpha-glucosidase (GAA). Normally, GAA is used by the body's cells to break down glycogen (a stored form of sugar) within specialized structures called lysosomes. In patients with Pompe disease, an excessive amount of glycogen accumulates and is stored in various tissues, especially heart and skeletal muscle, which prevents their normal function.

This study is being conducted to collect prospective, observational data on patients with late-onset Pompe disease. Approximately 60 subjects with late-onset Pompe disease will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* The patient must provide signed, informed consent prior to performing any study-related procedures.
* The patient must have a diagnosis of Pompe disease based upon: a) documented marked deficiency of GAA activity by muscle biopsy, skin fibroblasts, or leukocytes OR b) documented GAA gene mutation by deoxyribonucleic acid (DNA) analysis
* The patient must be greater than 8 years of age if enrolled at a site in the U.S. and greater than 18 years of age if enrolled at a site in Europe
* The patient must have documented onset of symptoms of Pompe disease after 12 months of age
* The patient must have at least 3 testable muscle groups in the arms and 3 testable muscle groups in the legs using quantitative muscle testing
* The patient must be able to perform pulmonary and muscle function testing in the supine position
* The patient must be able to provide reproducible muscle and pulmonary function test results within 10% of each other performed on Day 1 and Day 2 of the Screening/Baseline visit and forced vital capacity measurements within 10% of each other performed in the upright position on Day 1 and Day 2 of the Screening/Baseline visit
* The patient must have the ability to comply with the clinical protocol

Exclusion Criteria:

* The patient is unable to ambulate (use of assistive devices, such as walker, cane, crutches, is permitted);
* The patient requires the use of invasive ventilatory support.
* The patient requires the use of noninvasive ventilatory support during waking hours.
* The patient has received enzyme replacement therapy with acid alpha-glucosidase from any source
* The patient has received an investigational drug within 30 days prior to study enrollment, or is currently enrolled in another study which involves clinical evaluations
* The patient has a medical condition, serious intercurrent illness, or other extenuating circumstance that, in the opinion of the Investigator, may significantly interfere with study compliance including all prescribed evaluations and follow-up activities
* The patient has a major congenital abnormality
* For female patients only, the patient is pregnant or lactating, or is unwilling to practice birth control methods during the course of the study

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Late-Onset Patients diagnosed with Pompe Disease
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2004-03; Primary Completion 2005-05 (Actual); Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (5):
- United States (3):
  - Children's Hospital Medical Center, Washington D.C., District of Columbia
  - School of Medicine, Campus Box 8111, St Louis, Missouri
  - Children's Hospital & Regional Medical Center, Seattle, Washington
- Institut de Myologie, Groupe Hospitalier Pitie-Salpetriere, Batimant Babinski, Paris, France
- Universitair Medisch Centrum, Utrecht, Netherlands